CLINICAL TRIAL: NCT04885686
Title: Endodontic Post-operative Pain Evaluation of Patients After Using Endomethasone N or Endomethasone SP Root Canal Sealer: a Prospective, Comparative Randomized Clinical Trial
Brief Title: Endodontic Post-operative Pain Evaluation of Patients After Using Endomethasone N or Endomethasone SP (EndoPOP)
Acronym: EndoPOP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Septodont (Industry)
Collaborators: Slb Pharma (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EndoPOP; 2021-A00065-36 (Other: [French National Agency of Medicines and Health products])
Record Dates: First submitted 2021-04-29; First posted 2021-05-13 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-04

CONDITIONS: Root Canal Obturation
Keywords: Endodontics; root canal sealer; post-operative pain; zinc oxide eugenol; hydrocortisone; corticoid; root canal treatment
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Intervention Model Description: Study subject will be randomized in a 1:1 allocation ratio between the 2 treatment groups; the allocation will be stratified by pre-operative pain (3 classes) and center (12 classes).
Who Masked: Participant
Masking Description: The color of the two powders are not the same. The dentist will not be blinded to the treatment, but the patient will. The study is simple-blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Endomethasone N RCS (Experimental): Endomethasone N RCS is used in combination with gutta percha points for the permanent obturation of root canals.
  Interventions: Device: Endomethasone N RCS
- Endomethasone SP RCS (Active Comparator): Endomethasone SP RCS is used in combination with gutta percha points for the permanent obturation of root canals.
  Interventions: Device: Endomethasone SP RCS

INTERVENTIONS:
Device: Endomethasone N RCS — Root canal sealer
  Arms: Endomethasone N RCS
Device: Endomethasone SP RCS — Root canal sealer
  Arms: Endomethasone SP RCS

SUMMARY:
The study is a post-marketing performance and safety study, designed as a comparative, prospective, multicenter, simple-blind, randomized clinical trial. 300 subjects requiring a primary or a secondary root canal treatment will be enrolled in 2 groups (150 in each group). The aim of the study is to demonstrate the superiority of the hydrocortisone-containing root canal sealer Endomethasone N RCS, compared to the hydrocortisone-free root canal sealer Endomethasone SP RCS, with regard to reduction of the maximum post-operative spontaneous pain during the 7 days following the root canal treatment.

Root canal treatment procedures will be in accordance with the allocation by randomisation of Endomethasone N RCS or Endomethasone SP RCS. The spontaneous and the Masticatory pain will be record at predefined times, a phone call will be done at 48h and a visit will be realized at day 7 (max Day 14).

ELIGIBILITY:
Inclusion Criteria:

* Adult male or female (age ≥ 18 years);
* Patient requiring root canal treatment or retreatment;
* Patient who will need a single visit for the root canal therapy, for a mature molar or second premolar, with or without pre-operative pain
* Patient who received information and gave written consent (signed informed consent form);
* Subject affiliated to a health insurance system, or is a beneficiary (art. L.1121-11, Code of Public Health, France).

Exclusion Criteria:

* Pulpotomy or pulpectomy performed at a prior visit;
* Tooth with apical calcification (sealer unable to reach the root apex);
* Tooth with suspected root perforation;
* Immature tooth (too wide root apex requiring an apexification);
* Other dental treatment ongoing or scheduled within the study period;
* At least one symptomatic tooth among those that are not included in this study
* Known hypersensitivity to steroids, local anesthetics, or any component of study medical devices;
* Subject using long term anti-inflammatory drugs;
* Use of illicit substances during the 48h before the first visit (cannabis, cocaine…);
* Presence of any significant medical finding or significant history such as uncontrolled systemic diseases that may impact the safety, the interpretation of the results and/or the participation of the subject in the study according to the opinion of the investigator;
* Subject who cannot be contacted in case of emergency (phone number);
* Simultaneous participation in another clinical trial or subject still within the exclusion period of a previous clinical trial;
* Vulnerable subjects (art. L.1121-5 and L.1122-1-2, Code of Public Health, France; art. 66 of the Regulation (EU) 2017/745 on medical devices)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2021-06-22 (Actual); Primary Completion 2021-07-06 (Actual); Study Completion 2022-06-11 (Actual)

PRIMARY OUTCOMES:
Maximum post-operative pain using a visual analogue scale (VAS : 0-100) | from the end of the root canal treatment (Day 0) to Day 7
  The pain is assessed by patients in a diary using a Visual Analogue Scale (VAS: 0-100 mm; 0 no pain - 100 maximum pain) at different times after endodontic treatment (at the end of the root canal obturation, 3h, 6h 12h, 24h, Day 2, Day 3, Day 4 Day 5, Day 5, Day 7). The maximum pain felt will be compared between the 2 groups.

SECONDARY OUTCOMES:
Spontaneous pain intensity | from the end of the root canal treatment (Day 0) to Day 7
  The spontaneous pain intensity measured using a Visual Analogue Scale (VAS: 0-100mm; 0 no pain - 100 maximum pain)
Occurrence of spontaneous pain flare-ups | From Day 3 to Day7
  The occurrence of spontaneous pain flare-ups is an increase of 20 mm in the Visual Analogue Scale (VAS: 0-100mm; 0 no pain-100 maximum pain) between 2 consecutive measurements after the firsts 3 days.
Masticatory pain intensity | from the end of the root canal treatment (Day 0) to Day 7
  The masticatory pain intensity measured using a Visual Analogue Scale (VAS: 0-100mm; 0 no pain -100 maximum pain) assessed twice a day from Day 0 to Day3 (lunch and dinner), and once a day from Day 4 to Day7 (dinner).
Maximum Masticatory pain intensity using a visual analogue scale (VAS : 0-100mm) | from the end of the root canal treatment (Day 0) to Day 7
  The maximum masticatory pain intensity measured Visual Analogue Scale (VAS: 0-100mm; 0 no pain- 100 maximum pain)
Use of oral pain treatment | from the end of the root canal treatment (Day 0) to Day 7
  Patients reported the consumption of analgesic treatment in a diary. The proportion of patients who took oral pain medication and the treatment categories will be compared between the 2 groups.
Quality of life with the OHIP-17 questionnaire (score 0-68) | baseline and from 48 to 72 hours
  The answers and the total score from the OHIP 17-items questionnaire (measured at baseline and 48 h) will be compared between 2 groups. Score between 0 and 68, 0 means no dental issuel, 68 all the issues very often.
Adverse events | from the inclusion (Day 0) to Day 7
  Adverse events reported by patients on a diary from Day 0 to Day 7 and adverse events clinically observed by the dental surgeon at each follow-up visit will be used to assess the safety of root canal sealers and endodontic procedures

CONTACTS AND LOCATIONS:
Overall Officials: Yves BOUCHER, PU-PH, Study Director — APHP
Locations (15):
- France (15):
  - Cabinet dentaire, Agon-Coutainville
  - Cabinet dentaire, Betton
  - Cabinet dentaire, Chartres-de-Bretagne
  - Cabinet Dentaire, Cherbourg
  - Cabinet dentaire, Cherbourg
  - Cabinet dentaire, Dinan
  - Cabinet dentaire, Équeurdreville-Hainneville
  - Cabinet dentaire, Lamballe
  - Centre de santé dentaire Chevaleret, Paris
  - Centre dentaire Flandre, Paris
  - Cabinet dentaire, Pluguffan
  - Cabinet dentaire, Quimper
  - Cabinet dentaire, Rennes
  - Cabinet dentaire, Saint-Aubin-de-Médoc
  - Cabinet dentaire, Tinténiac

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Boucher Y, Abrgall H, Bar V, Basl-Th Bault FO, Cano S, Colombel H, Le Guicher G, Cameli C. Spontaneous and Masticatory Post-endodontic Pain After Using Endomethasone N vs SP Root Canal Sealers: A Randomised Controlled Clinical Trial. Eur Endod J. 2024 Aug 22;9(3):218-230. doi: 10.14744/eej.2024.96977. PMID 38644670